CLINICAL TRIAL: NCT03382496
Title: EVIDENS: Lung Cancer Patients Treated With Nivolumab: A Longitudinal, Prospective, Observational, Multicentric Study
Brief Title: Observational Study for Lung Cancer Patients Treated With Nivolumab
Acronym: EVIDENS
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-417
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung Cancer patients in France: Lung Cancer patients treated by nivolumab in real life condition in France from October 2016 to October 2017
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
This study will describe the characteristics of patients initiating nivolumab treatment for lung cancer and their outcomes over 3 years in France

ELIGIBILITY:
Inclusion Criteria:

* Male or female: 18 age at the time of nivolumab initiation
* Pathologically confirmed diagnosis of lung cancer
* Patient initiating nivolumab :therapeutic decision to initiate nivolumab must be taken by the physician prior to enrolling a patient in the study

Exclusion Criteria:

-Patient taking part in an interventional study for lung cancer treatment for which nivolumab is 1 of the investigational drugs

Other protocol defined inclusion or exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to collect data for patients diagnosed with a lung cancer and initiating nivolumab in France
Sampling Method: Non-Probability Sample
Enrollment: 1462 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Distribution of gender | At baseline
Distribution of age | At baseline
Distribution of line of therapy at nivolumab initiation | At baseline
Distribution of ECOG PS | At baseline
  Eastern Cooperative Oncology Group Performance Status (ECOG PS) A scale used to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis
Distribution of patients working status at nivolumab initiation | At baseline
QoL (EQ-5D) at nivolumab initiation | At baseline
  Quality of Life (QoL) as assessed by European Quality of Life-5 Dimensions (EQ-5D) EQ-5D: the descriptive system consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with 3 levels (eg, no problems, moderate problems, extreme problems)
Median time from initial diagnosis to nivolumab initiation | At baseline
  Median time from initial diagnosis to nivolumab initiation (derived from date of initial diagnosis and date of first dose of nivolumab, assumed to be the date of D0 visit). Any lung cancer declaring more than 5 years after another cancer is defined as an initial diagnosis of lung cancer
Number of patients exposed to other lung cancer treatments | At baseline
Distribution of current smokers, former smokers, and non-smokers at initial diagnosis | At baseline
Distribution of cancer stage at initial diagnosis and at nivolumab initiation | At baseline
Distribution of Lung cancer histology at initial diagnosis | At baseline
Number of patients with untreated brain metastasis at nivolumab initiation | At baseline
Number of patients with treated brain metastasis at nivolumab initiation | At baseline
Number of patients with PD-L1 expression at nivolumab initiation | At baseline
  PD-LI (Programmed death-ligand 1)
Number of patients with mutations at nivolumab initiation | At baseline
Distribution of concomitant diseases at nivolumab initiation | At baseline
Number of patients with corticosteroids treatment at nivolumab initiation | At baseline
(OS) Overall Survival | Up to 3 years
  Time from index date (treatment with nivolumab) until date of death due to any cause

SECONDARY OUTCOMES:
Overall Survival after initiation of nivolumab | Up to 2 years
Distribution of nivolumab adverse drug reaction | At 3 years after nivolumab initiation
Progression Free Survival (PFS) | Up to 3 years after nivolumab initiation
  PFS measured by time since index date (initial treatment with nivolumab) to either the first disease progression date or last known tumor assessment date, or death due to any cause, whichever occurs first as assessed by RECIST 1.1
Objective Response Rate (ORR) | Up to 3 years after nivolumab initiation
  ORR is measured by the sum of partial responses plus complete responses as assessed by (RECIST 1.1) Response Evaluation Criteria In Solid Tumors
Quality of Life (QoL) | Baseline to 3 years after nivolumab initiation
Distribution of patient management treatment patterns | Baseline to 3 years
Mean weight change in kilogram from baseline | Baseline up to 3 years
Mean ECOG PS change from baseline | Baseline up to 3 years
Distribution of patients with new metastasis | Up to 3 years
Distribution of patients with progression of pre-existing sites | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Fontaine-lès-Dijon, France

REFERENCES:
- [Derived] Barlesi F, Dixmier A, Debieuvre D, Raspaud C, Auliac JB, Benoit N, Bombaron P, Moro-Sibilot D, Audigier-Valette C, Asselain B, Egenod T, Rabeau A, Fayette J, Sanchez ML, Labourey JL, Westeel V, Lamoureux P, Cotte FE, Allan V, Daumont M, Dumanoir J, Reynaud D, Calvet CY, Ozan N, Perol M. Effectiveness and safety of nivolumab in the treatment of lung cancer patients in France: preliminary results from the real-world EVIDENS study. Oncoimmunology. 2020 Apr 12;9(1):1744898. doi: 10.1080/2162402X.2020.1744898. PMID 33457089
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html